CLINICAL TRIAL: NCT02769494
Title: The Efficacy of Topically Applied Mesalazine Sustained-Release Tablets in Oral Lesions of Crohn's Disease
Brief Title: The Efficacy of Topical Mesalazine Sustained-Release Tablets in Crohn's Disease Patients With Oral Ulcer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Doctor of Xijing Hospital of Digestive Diseases,Principal, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20160107-1
Record Dates: First submitted 2016-03-09; First posted 2016-05-11 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Crohn's Disease; Oral Ulcer
Keywords: Oral ulcer; Crohn's disease
MeSH Terms: conditions — Crohn Disease; Oral Ulcer | interventions — Mesalamine; Flavin Mononucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesalazine Group (Experimental): Mesalazine Sustained-Release Tablets and 0.02L glycerol mixed, 2.5% mesalazine glycerol suspension liquid, gently apply to the ulcer surface, 3 times/day. Daily treatment time of the drug is 8 am,12 pm and 4 pm.
  Interventions: Drug: Mesalazine Sustained-Release Tablets
- Riboflavin Sodium Phosphate Group (Active Comparator): wipe the riboflavin sodium phosphate injection to the ulcer surface, 3 times/day. Daily treatment time of the drug is am,12 pm and 4 pm.
  Interventions: Drug: Riboflavin Sodium Phosphate Injection

INTERVENTIONS:
Drug: Mesalazine Sustained-Release Tablets — Mesalazine sustained-release tablets 500mg and 0.02L glycerol mixed, the preparation of 2.5% the mesalazine glycerol suspension liquid, gently apply to the ulcer surface, 3 times/day. The application time of the drug is 8:00,12:00, 16:00. Daily 20:00 measure the size of the mouth ulcers and record the symptoms in the diary card.
  Other Names: Pentasa
  Arms: Mesalazine Group
Drug: Riboflavin Sodium Phosphate Injection — gently apply the riboflavin sodium phosphate injection to the ulcer surface, 3 times/day. The application time of the drug is 8:00,12:00, 16:00. Daily 20:00 measure the size of the mouth ulcers and record the symptoms in the diary card.
  Arms: Riboflavin Sodium Phosphate Group

SUMMARY:
This study aims at evaluating efficacy and safety of topical using Mesalazine Sustained-Release Tablets in in the treatment of oral ulcers in patients with Crohn's disease.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up.

Screening: This phase will last a maximum of 7 days and subjects eligibility will be evaluated after informed consent signature.

Treatment: Subjects are randomly assigned to treatment and will be treated for 7 days. Daily oral ulcer area and symptoms were recorded during the treatment period. A randomization visit will take place on day 0 and an end-of-treatment visit will take place between day 6 and 8.

Follow-up: 28 days after the end of treatment. Efficacy of treatment was evaluated by the oral ulcer remission or decreasing.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~65, both gender.
* Patients with oral ulcer and confirmed Crohn's disease.

Exclusion Criteria:

* Contraindications to study drugs.
* Underwent or will accept oral Surgery.
* Patients are not able to sign the informed consent or not comply with the study protocol.
* Planning for pregnancy, pregnancy and lactating women.
* Enrolled in other clinical trials in the past 30 days.
* Patients with concurrent / new other serious diseases will affect the effectiveness and safety evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
oral ulcer healing | the 7 Days of treatment.
  The primary outcome is ulcer healing, oral ulcer area can be divided into 3 degrees: 1 degrees for a single ulcer, area ≤ 8mm; 2 degree for a single ulcer, 8mm ≤ area ≤ 15mm, or two ulcers, area of every ulcer ≤ 8mm; 3 degree for a single ulcer, area ≥ 15 mm, or 2 ulcers, every area between 8 to 15mm. Recovery refers oral ulcer is healing completely. The effective is the ulcer area decrease more than 1 degree. Invalid means the ulcer area is no change.
oral ulcer recurrence | the 28 Days after the end of treatment.
  to observe the recurrence rate of ulcer

SECONDARY OUTCOMES:
symptoms effective rates | At the 7 Days of the treatment, and the 28 Days after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%. Total score = frequency + severity. Frequency score is calculated by all the frequency of oral pain, anorexia,and eating difficult. Severity is accumulated by the degree of symptoms described above,which is divided to 4 degree as 0 presenting none,and 3 presenting most severe.
adverse events | From 1st Day to 7th Days of the treatment and the 28 Days after the end of treatment.
  Participants with Adverse Events as a Measure of Safety and Tolerability. The common side effects of the study include headache, diarrhea, nausea, abdominal pain, vomiting and skin rash.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, Ph. D, Study Director — Degistive Disease of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No